CLINICAL TRIAL: NCT03746522
Title: A Phase 3 Trial of Setmelanotide (RM-493), a Melanocortin-4 Receptor (MC4R) Agonist, in Bardet-Biedl Syndrome (BBS) and Alström Syndrome (AS) Patients With Moderate to Severe Obesity
Brief Title: Setmelanotide (RM-493), Melanocortin-4 Receptor (MC4R) Agonist, in Bardet-Biedl Syndrome (BBS) and Alström Syndrome (AS) Participants With Moderate to Severe Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM-493-023; 2018-004058-11 (EudraCT Number)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bardet Biedl Syndrome (BBS); Alström Syndrome (AS)
Keywords: MC4R Pathway; Obesity; BBS; AS
MeSH Terms: conditions — Bardet-Biedl Syndrome; Alstrom Syndrome; Obesity | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Setmelanotide (Double-Blind) (Experimental): Participants received once daily SC injection of setmelanotide for 14 weeks in a double-blind placebo-controlled treatment period (Period 1). Participants ≥16 years of age started on setmelanotide 2.0 mg with dose escalation to 3.0 mg. Participants <16 years of age started on setmelanotide 1.0 mg with dose escalation to 3.0 mg.
  Interventions: Drug: Setmelanotide
- Placebo (Double-Blind) (Placebo Comparator): Participants received once daily SC injection of placebo (matching setmelanotide) for 14 weeks in a double-blind placebo-controlled treatment period (Period 1).
  Interventions: Drug: Placebo
- Setmelanotide (Open-label) (Experimental): After the initial 14-week double-blind treatment period, all participants immediately transitioned to open-label setmelanotide once daily SC injection for 38 weeks (Period 2) and then continued to receive setmelanotide in the 14-week open-label treatment period (Period 3).
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — SC injection of setmelanotide
  Other Names: SET; RM-493
  Arms: Setmelanotide (Double-Blind); Setmelanotide (Open-label)
Drug: Placebo — SC injection of placebo
  Arms: Placebo (Double-Blind)

SUMMARY:
This pivotal, phase 3 study is designed to confirm the efficacy and safety of setmelanotide, a potent melanocortin receptor type 4 (MC4R) agonist, for the treatment of obesity and hyperphagia in participants with Bardet Biedl syndrome (BBS) or Alström syndrome (AS). The study's primary efficacy endpoint is to evaluate the proportion of participants (≥ 12 years of age at baseline) who lose ≥ 10% of their baseline body weight following approximately (~) 52 weeks of treatment with setmelanotide compared to a historical control rate.

DETAILED DESCRIPTION:
Eligible participants will enter a 14-week, randomized, double-blind, placebo-controlled treatment period (Period 1) that will be followed by a 38-week open-label treatment period (Period 2) in which all participants will receive setmelanotide. Following Period 2, participants will continue receiving open-label setmelanotide for 14 weeks (Period 3), after which they could enroll into a separate treatment extension study.

ELIGIBILITY:
Inclusion Criteria:

1. BBS clinical diagnosis or AS diagnosis
2. Greater than or equal to (≥) 6 years of age.
3. Obese, defined as BMI ≥30 kilograms/meters^2 for participants ≥16 years of age or weight >97th percentile for age and sex on growth chart assessment for participants 6 to 15 years of age.
4. Study participant and/or parent or guardian is able to communicate well with the Investigator, to understand and comply with the requirements of the study, and is able to understand and sign the written informed consent/assent.
5. Female participants of child-bearing potential must be confirmed non-pregnant and agree to use contraception as outlined in the protocol. Female participants of non-childbearing potential, defined as: surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation), post-menopausal for at least 12 months (and confirmed with a screening follicle stimulating hormone (FSH) level in the post-menopausal lab range), or failure to have progressed to Tanner Stage V and/or failure to have achieved menarche, do not require contraception during the study.
6. Male participants with female partners of childbearing potential must agree to use a double barrier method contraception if they become sexually active during the study or within 90 days following their participation in the study. Male participants must also not donate sperm during and for 90 days following their participation in the study.

Exclusion Criteria:

1. Recent intensive (within 2 months) diet and/or exercise regimen with or without the use of weight loss agents (including herbal medications) that has resulted in >2% weight loss. These participants may be reconsidered approximately 1 month after cessation of such intensive regimens.
2. Current or prior (within prior 2 months) use of any medication, including those approved to treat obesity, that could impact the efficacy results of this study (e.g., orlistat, lorcaserin, phentermine-topiramate, naltrexone-bupropion, liraglutide). Participants on a stable dose and regimen (for at least 2 months) of medication to treat attention deficit hyperactivity disorder (ADHD) may be enrolled in the study as long as they agree to remain on the same dose and regimen during the study.
3. Prior gastric bypass surgery resulting in >10% weight loss durably maintained from the baseline pre-operative weight with no evidence of weight regain. Specifically, participants may be considered if surgery was not successful, resulted in <10% weight loss compared to pre-operative baseline weight, or there is clear evidence of weight regain after an initial response to bariatric surgery. All participants with a history of bariatric surgery must be discussed with, and receive approval from, the Sponsor prior to enrollment.
4. Diagnosis of schizophrenia, bipolar disorder, personality disorder or other Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-V) disorders that the Investigator believes will interfere significantly with study compliance. Neurocognitive disorders affecting ability to consent will not be disqualifying as long as an appropriate guardian able to give consent has been appointed.
5. In participants with no significant neurocognitive deficits:

   * A Patient Health Questionnaire-9 (PHQ-9) score of ≥15 and/or
   * Any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS), any lifetime history of a suicide attempt, or any suicidal behavior in the last month.
6. Current, clinically significant pulmonary, cardiac, or oncologic disease considered severe enough to interfere with the study and/or confound the results. Any participant with a potentially clinically significant disease should be reviewed with the Sponsor to determine eligibility.
7. History of significant liver disease or liver injury, or a current liver assessment due to abnormal liver tests (as indicated by abnormal liver function tests, alanine transaminase [ALT], aspartate transaminase [AST], alkaline phosphatase, or serum bilirubin >1.5x the upper limit of normal [ULN] for any of these tests) for an etiology other than non-alcoholic fatty liver disease (NAFLD). Thus, any underlying etiology besides NAFLD, including diagnosed non-alcoholic steatohepatitis (NASH), other causes of hepatitis, or history of hepatic cirrhosis is exclusionary, but the presence of NAFLD is not exclusionary.
8. Moderate to severe renal dysfunction defined as <30 mL/min.
9. History or close family history (parents or siblings) of skin cancer or melanoma (excluding non-invasive basal or squamous cell lesion), or participant history of ocular-cutaneous albinism.
10. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions (excluding non-invasive basal or squamous cell lesion).
11. Participant is, in the opinion of the Study Investigator, not suitable to participate in the study.
12. Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
13. Significant hypersensitivity to study drug.
14. Inability to comply with once daily (QD) injection regimen.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (12):
- United States (6):
  - Wr-McCr, Llc, San Diego, California
  - UMMS Baystate Health; BAYSTATE MEDICAL CENTER; Baystate Children's Specialty Center, Springfield, Massachusetts
  - Columbia University Center, New York, New York
  - M3 Wake Research, Raleigh, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Alberta Health Services, Edmonton, Alberta, Canada
- France (2):
  - Sorbonne University, Hôpital de la Pitié-Salpêtrière, Paris
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
- UPR Medical Sciences Campus, Rio Piedras, Puerto Rico
- Universidad Autónoma de Madrid University Hospital Niño, Madrid, Spain
- St. Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ervin C, Norcross L, Mallya UG, Fehnel S, Mittleman RS, Webster M, Haqq AM, Haws RM. Interview-Based Patient- and Caregiver-Reported Experiences of Hunger and Improved Quality of Life with Setmelanotide Treatment in Bardet-Biedl Syndrome. Adv Ther. 2023 May;40(5):2394-2411. doi: 10.1007/s12325-023-02443-y. Epub 2023 Mar 24. PMID 36961653
- [Derived] Forsythe E, Haws RM, Argente J, Beales P, Martos-Moreno GA, Dollfus H, Chirila C, Gnanasakthy A, Buckley BC, Mallya UG, Clement K, Haqq AM. Quality of life improvements following one year of setmelanotide in children and adult patients with Bardet-Biedl syndrome: phase 3 trial results. Orphanet J Rare Dis. 2023 Jan 16;18(1):12. doi: 10.1186/s13023-022-02602-4. PMID 36647077
- [Derived] Haqq AM, Chung WK, Dollfus H, Haws RM, Martos-Moreno GA, Poitou C, Yanovski JA, Mittleman RS, Yuan G, Forsythe E, Clement K, Argente J. Efficacy and safety of setmelanotide, a melanocortin-4 receptor agonist, in patients with Bardet-Biedl syndrome and Alstrom syndrome: a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial with an open-label period. Lancet Diabetes Endocrinol. 2022 Dec;10(12):859-868. doi: 10.1016/S2213-8587(22)00277-7. Epub 2022 Nov 7. PMID 36356613
- [Derived] Haws RM, Gordon G, Han JC, Yanovski JA, Yuan G, Stewart MW. The efficacy and safety of setmelanotide in individuals with Bardet-Biedl syndrome or Alstrom syndrome: Phase 3 trial design. Contemp Clin Trials Commun. 2021 May 3;22:100780. doi: 10.1016/j.conctc.2021.100780. eCollection 2021 Jun. PMID 34013094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in pivotal cohort (38 participants) or supplemental cohort (14 participants) and received setmelanotide/placebo for the 14-week double-blind period (Period 1) followed by setmelanotide in the open-label period (Period 2 and 3).
Pre-assignment Details: As planned, the analysis of the primary and secondary endpoints were done only in the pivotal cohort.
  Pivotal cohort: All the enrolled Bardet-Biedl syndrome (BBS)/Alström Syndrome (AS) participants at the time of the planned sixth AS participant enrollment.
  Supplemental cohort: Any additional participants enrolled were included in supplemental cohort.
Groups:
- Setmelanotide (Double-Blind): Participants received once daily subcutaneous (SC) injection of setmelanotide for 14 weeks in a double-blind placebo-controlled treatment period (Period 1). Participants ≥16 years of age started on setmelanotide 2.0 mg with dose escalation to 3.0 mg. Participants <16 years of age started on setmelanotide 1.0 mg with dose escalation to 3.0 mg.
Period: Period 1: Double-Blind (14 Weeks)
Arm/Group | Setmelanotide (Double-Blind) | Placebo (Double-Blind) | Setmelanotide (Open-label)
Started | 27 | 25 | 0
Completed | 27 | 23 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Period 2: Open-Label (38 Weeks)
Arm/Group | Setmelanotide (Double-Blind) | Placebo (Double-Blind) | Setmelanotide (Open-label)
Started | 0 | 0 | 50
Completed | 0 | 0 | 41
Not Completed | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Other than specified | 0 | 0 | 2
Period: Period 3: Open-Label (14 Weeks)
Arm/Group | Setmelanotide (Double-Blind) | Placebo (Double-Blind) | Setmelanotide (Open-label)
Started | 0 | 0 | 41
Completed | 0 | 0 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set defined as participants who received at least 1 dose of study drug (placebo or setmelanotide).
Groups:
- Setmelanotide: Participants received once daily SC injection of setmelanotide for 14 weeks in a double-blind placebo-controlled treatment period (Period 1). Participants ≥16 years of age started on setmelanotide 2.0 mg with dose escalation to 3.0 mg. Participants <16 years of age started on setmelanotide 1.0 mg with dose escalation to 3.0 mg. After the initial 14-week double-blind treatment period, all participants immediately transitioned to open-label setmelanotide once daily SC injection for 38 weeks (Period 2) and then continued to receive setmelanotide in the 14-week open-label treatment period (Period 3).
- Placebo: Participants received once daily SC injection of placebo (matching setmelanotide) for 14 weeks in a double-blind placebo-controlled treatment period (Period 1). After the initial 14-week double-blind treatment period, all participants immediately transitioned to open-label setmelanotide once daily SC injection for 38 weeks (Period 2) and then continued to receive setmelanotide in the 14-week open-label treatment period (Period 3).
- Total: Total of all reporting groups
Arm/Group | Setmelanotide | Placebo | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (9.95) | 20.7 (12.05) | 19.5 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 14 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 21 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 4 | 3 | 7
  United States | 16 | 17 | 33
  United Kingdom | 0 | 2 | 2
  France | 4 | 1 | 5
  Spain | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (≥12 Years of Age at Baseline) Who Reached ≥10% Weight Loss Threshold After 1 Year (Period 2): Pivotal Cohort
Description: The percentage of participants (≥12 years of age at baseline) who achieved a ≥10% reduction from baseline in body weight at Period 2 or after 52 weeks of treatment with setmelanotide were analyzed. There was a 14-week placebo-controlled period at the beginning of the trial. After completion of the placebo-controlled period, all participants from the placebo group switched to setmelanotide treatment. The placebo group was integrated into the 52-week analysis so that the participants who received placebo, had 52 weeks of setmelanotide treatment after the first dose of "active" treatment. Placebo participants were also included in this analysis.
Time Frame: 52 weeks
Population: Participants in the Full Analysis Set (defined as randomized participants who received at least 1 dose of study drug and had active treatment baseline [ATB] data) with available data were analyzed. Participants in the pivotal cohort who received setmelanotide (and were ≥12 years of age) were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pivotal Cohort: Participants received once daily SC injection of setmelanotide/placebo for 14 weeks in a double-blind placebo-controlled treatment period (Period 1). After the initial 14-week double-blind treatment period, all participants immediately transitioned to open-label setmelanotide once daily SC injection for 38 weeks (Period 2).
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 31
percentage of participants | 32.3 [16.7 to 51.4]
Statistical Analysis 1: Comparison: Pivotal Cohort; Test type: Other; p = 0.0006, Rubin's Rule — P-value was one-sided and compared with alpha = 0.025

2. Secondary Outcome: Mean Percent Change From Baseline in Body Weight (≥12 Years of Age) at Week 52 (Period 2): Pivotal Cohort
Description: The mean percent change from baseline in body weight at 52 weeks was analyzed. There was a 14-week placebo-controlled period at the beginning of the trial. After completion of the placebo-controlled period, all participants from the placebo group switched to setmelanotide treatment. The placebo group was integrated into the 52-week analysis so that the participants who received placebo, had 52 weeks of setmelanotide treatment after the first dose of "active" treatment. Placebo participants were also included in this analysis.
Time Frame: Baseline, Week 52
Population: Participants in the Full Analysis Set with available data were analyzed. Participants in pivotal cohort who received setmelanotide (and were ≥12 years of age) were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 31
percent change | -5.21 (7.895)
Statistical Analysis 1: Comparison: Pivotal Cohort; Test type: Other; p = 0.0005, Rubin's Rule — p-value was one-sided and compared with alpha = 0.025

3. Secondary Outcome: Mean Percent Change From Baseline in the Weekly Average of the Daily Hunger Score (≥12 Years of Age) at Week 52 (Period 2): Pivotal Cohort
Description: Mean percent change in hunger scores for participants ≥12 years of age with leptin receptor (LEPR) deficiency obesity in treatment with setmelanotide was evaluated. Hunger score ranged from 0= "not hungry at all" to 10= "hungriest possible" on Likert-type scale. On Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on weekly basis. Weekly average hunger score of daily worst (most) hunger score in 24 hours is the hunger score used to assess this study endpoint. There was a 14-week placebo-controlled period at the beginning of the trial. After completion of the placebo-controlled period, all participants from the placebo group switched to setmelanotide treatment. Placebo group was integrated into the 52-week analysis so that participants who received placebo, had 52 weeks of setmelanotide treatment after the first dose of "active" treatment. Placebo participants were also included in this analysis.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 16
percent change | -30.91 (24.733)
Statistical Analysis 1: Comparison: Pivotal Cohort; Test type: Other; p < 0.0001, Rubin's Rule — p-value was one-sided and compared with alpha=0.025

4. Secondary Outcome: Number of Participants (≥12 Years of Age With no Cognitive Impairment) Who Achieved a ≥ 25% Improvement in the Weekly Average of the Daily Hunger Score From Baseline at Week 52 (Period 2): Pivotal Cohort
Description: Number of participants (≥12 years of age with no cognitive impairment) achieving ≥25% improvement from baseline in hunger score at Week 52 was assessed. Hunger score ranged from 0= "not hungry at all" to 10= "hungriest possible" on Likert-type scale. On Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on weekly basis. Weekly average hunger score of daily worst (most) hunger score in 24 hours is the hunger score used to assess this study endpoint. There was a 14-week placebo-controlled period at the beginning of the trial. After completion of placebo-controlled period, all participants from placebo group switched to setmelanotide treatment. Placebo group was integrated into the 52-week analysis so that participants who received placebo, had 52 weeks of setmelanotide treatment after the first dose of "active" treatment. Placebo participants were also included in this analysis.
Time Frame: Baseline, Week 52
Population: Participants in Full Analysis Set with available data were analyzed. Participants in pivotal cohort who received setmelanotide (and were ≥12 years of age) were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal Cohort
Number analyzed (Participants) | 16
Participants | 10
Statistical Analysis 1: Comparison: Pivotal Cohort; Test type: Other; p < 0.0001, Rubin's Rule — p-value was one-sided and compared with alpha = 0.025

ADVERSE EVENTS:
Time Frame: Double-blind: From first dose up to Week 14 Open-label: From Week 14 up to Week 66
Description: Safety Analysis Set was defined as participants who received at least 1 dose of study drug (placebo or setmelanotide). Participants in the pivotal and supplemental cohorts were included.
Groups:
- Setmelanotide (Double-Blind Period): Participants received once daily SC injection of setmelanotide for 14 weeks in a double-blind placebo-controlled treatment period (Period 1).
- Placebo (Double-Blind Period): Participants received once daily SC injection of placebo (matching setmelanotide) for 14 weeks in a double-blind placebo-controlled treatment period (Period 1).
Arm/Group | Setmelanotide (Double-Blind Period) | Placebo (Double-Blind Period) | Setmelanotide (Open-label)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/27 | 2/25 | 0/50
Other Adverse Events (participants affected / at risk) | 26/27 | 24/25 | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide (Double-Blind Period) (N=27) | Placebo (Double-Blind Period) (N=25) | Setmelanotide (Open-label) (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide (Double-Blind Period) (N=27) | Placebo (Double-Blind Period) (N=25) | Setmelanotide (Open-label) (N=50)
High density lipoprotein decreased (Investigations) | 4 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 6 | 7
Dizziness (Nervous system disorders) | 1 | 2 | 1
Injection site erythema (General disorders) | 12 | 11 | 4
Injection site pruritus (General disorders) | 8 | 9 | 4
Injection site pain (General disorders) | 3 | 8 | 5
Injection site bruising (General disorders) | 6 | 9 | 3
Injection site induration (General disorders) | 6 | 4 | 5
Fatigue (General disorders) | 1 | 2 | 3
Injection site haemorrhage (General disorders) | 3 | 2 | 1
Injection site oedema (General disorders) | 2 | 1 | 3
Injection site reaction (General disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 6 | 8
Vomiting (Gastrointestinal disorders) | 7 | 0 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3
Spontaneous penile erection (Reproductive system and breast disorders) | 1 | 0 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 17 | 0 | 19
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT03746522/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT03746522/SAP_001.pdf